CLINICAL TRIAL: NCT06541769
Title: CIPN-prevention Trial Evaluating the Efficacy of Hand-cooling and Hand-compression in Patients Undergoing (Neo-) Adjuvant Chemotherapy for Primary Breast Cancer
Brief Title: CIPN-prevention Trial Evaluating the Efficacy of Hand-cooling and Hand-compression
Acronym: POLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Laura Michel, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT/HD_GYNONC:POLAR
Record Dates: First submitted 2024-07-15; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Onychodystrophy
Keywords: Breast cancer; CIPN; Peripheral neuropathy; hypothermia
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Hypothermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermia (Experimental): limb Hypothermia with special hypothermia-gel-gloves of the dominant hand starting 30min before chemotherapy application and ending 30min after. The glove will be changed every 30min to provide constant cooling
  Interventions: Device: Limb hypothermia
- Compression (Experimental): compression of the dominant hand provided by one-way latex-gloves. The necessary size will be determined after measurement for every Patient individually
  Interventions: Device: Limb compression

INTERVENTIONS:
Device: Limb hypothermia — Limb hypothermia with special gel-gloves
  Arms: Hypothermia
Device: Limb compression — compression with sterile one way Latex gloves. Size measured for every Patient individually
  Arms: Compression

SUMMARY:
The POLAR study is a monocentric, prospective, randomized, 2-arm study designed to evaluate the effectiveness of compression or hypothermia in preventing higher-grade chemotherapy-induced peripheral neuropathy (CIPN) (Grade > 1 according to EORTC) in patients undergoing (neo-)adjuvant chemotherapy with weekly Paclitaxel or Nab-Paclitaxel. In this study, the dominant hand of participants will be either cooled or compressed, while the contralateral hand will serve as a control. The treatment groups will be randomized.

The primary aim of the study is to compare the effectiveness of limb hypothermia versus compression in preventing CIPN. Additionally, the investigators will assess the quality of life and therapy acceptance among the participants in both study arms. Data from the two groups will be collected and compared to determine the most effective intervention for preventing CIPN and to understand the overall impact on patients' well-being and treatment adherence.

DETAILED DESCRIPTION:
This is a prospective, randomized, two-arm study with the aim of assessing the effectiveness of compression or cooling in preventing higher-grade CIPN (>Grade 2 according to EORTC) during weekly paclitaxel or nab-paclitaxel based (neo-)adjuvant chemotherapy. For this purpose, the dominant hand is either cooled or compressed, depending on the study arm, and the contralateral hand is only observed. The allocation to compression or cooling is done through randomization. In a second step, the effectiveness of cooling should be compared with compression. For this purpose, the data collected from the two study arms will be compared. Furthermore, patient satisfaction and quality of life during therapy will be examined. The primary study endpoint is the difference in moderate and severe polyneuropathy (CTCAE grade ≥ 2) compared between the control hand and the intervention hand within the study arms (extremity with cooling vs. control extremity or extremity with compression vs. control extremity). CIPN is evaluated via CTCAE criteria 4.0 and by the Total Neuropathy Score (TNS; clinical version). In addition, sensorimotor symptoms are documented using EORTC QLQ-CIPN20 questionnaires (see also 3.3).

In a second, hierarchical test, the rate of moderate and severe polyneuropathies is compared between the two intervention arms (cooling vs. compression). The rate of onychodystrophies and onycholysis in both intervention arms (compression and cooling) is documented using CTAE criteria and compared between the intervention arm and the control arm as well as between both patient groups.

In addition, patient satisfaction and acceptance of the intervention are examined. EORTC QLQ-C30 questionnaires are used to document quality of life. Any toxicities during therapy are documented according to the CTCAE criteria 4.0.

ELIGIBILITY:
Inclusion Criteria:

- all female patients with signed informed consent who are starting with (neo-) adjuvant chemotherapy according to the following protocols:

* 4 x Epirubicin/Cyclophosphamid (EC) q3w, followed by 12 x Paclitaxel weekly or 12x Nab-Paclitaxel (+/- Trastuzumab)
* Paclitaxel or Nab-Paclitaxel weekly without anthracyclines
* Paclitaxel or Nab-Paclitaxel weekly in combination with Carboplatin

Exclusion criteria:

* patients without informed consent
* ECOG-Status > 1
* age under 18 years
* previous chemotherapy
* therapy with SSNRI, SSRI, or tricyclic antidepressants especially duloxetine, gabapentine, pregabaline and amitryptiline.
* known polyneuropathy (e.g. alcoholic PNP, nephrogenic PNP, diabetic PNP etc.)
* Patients having diseases connected to PNP:

  * Sjögren-syndrome, sarkoidosis, amyloidneuropathy, Morbus Fabry, HSAN (Hereditary Sensoric and Autonome Neuropathy)
  * Guillain-Barré-syndrome, acute intermittent porphyria, critical-illness-PNP
  * Vaskulitides, HNPP, diabetic amyotrophy, multifokal motoric neuropathy, Lewis-Sumner-syndrome, borreliosis-neuropathy, Zoster-neuritis, neuralgic shoulder amyotrophy
  * Myelopathy, compression of the myelon, syringomyelia, meningomyelitis, Restless-Legs-syndrome
  * Sulcus-Ulnaris-syndrome, Loge-de-Guyon-syndrome, Medianus-compression-syndrome, multiple sklerosis, AML, Lupus erythematodes, sklerodermia/systemic sclerosis, Ehlers-Danlos-syndrome, CREST-syndrome, Raynaud-syndrome, cold aglutinin disease, hämatologic neoplasms, diabetes mellitus, chronic alcohol abuse, hepatitis C, known severe kidney disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of CIPN grade >1 on the interventional hand compared to the non-interventional hand | 1 year (during taxane therapy and follow up)
  Comparing rates of CIPN>grade 1 on the interventional and non-interventional hand by evaluation CTCAE criteria, EORTC QLQ-CIPN-20, the clinical version of the total neuropathy score (TNSc), Magnetic resonance neurography (MRI; n=21) and nerve conduction studies (n=4)

SECONDARY OUTCOMES:
Incidence of onycholysis/onychodystrophy grade >1 on the interventional hand compared to the non-interventional hand | 1 year (during taxane therapy and follow up)
  Comparing rates of onycholysis/onychodystrophy>grade 1 on the interventional and non-interventional hand
Magnetic resonance neurography (MRI) as a possible marker of CIPN | 3 month (before and after taxane therapy)
  To evaluate the role of MRI as a possible marker for CIPN, MRI will be performed in a subset of patient (N=21)
Influence of CIPN on the quality of life | 1 year (during taxane therapy and follow up)
  Standardized clinical questionnaires (EORTC QLQ30, QLQ-CIPN-20) are used to determine the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Michel, M.D., Study Director — University Hospital Heidelberg
Locations (1):
- National Center for Tumor diseases (NCT), Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Michel LL, Schwarz D, Romar P, Feisst M, Hamberger D, Priester A, Kurre E, Klein E, Muller J, Schinkothe T, Weiler M, Smetanay K, Fremd C, Heublein S, Thewes V, Breckwoldt MO, Jager D, Bendszus M, Marme F, Schneeweiss A. Efficacy of Hand Cooling and Compression in Preventing Taxane-Induced Neuropathy: The POLAR Randomized Clinical Trial. JAMA Oncol. 2025 Apr 1;11(4):408-415. doi: 10.1001/jamaoncol.2025.0001. PMID 40048176